CLINICAL TRIAL: NCT00853658
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Active-controlled Study to Evaluate the Efficacy and Safety of Both Aliskiren Monotherapy and Aliskiren/Enalapril Combination Therapy Compared to Enalapril Monotherapy, on Morbidity and Mortality in Patients With Chronic Heart Failure (NYHA Class II - IV). The Study is Also Known as Aliskiren Trial of Minimizing OutcomeS in Patients With HEart Failure (ATMOSPHERE).
Brief Title: Efficacy and Safety of Aliskiren and Aliskiren/Enalapril Combination on Morbidity-mortality in Patients With Chronic Heart Failure
Acronym: ATMOSPHERE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100F2301; 2008-004104-31 (EudraCT Number)
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Cardiovascular death; CHF hospitalization; morbi-mortality trial; outcome study; endpoint driven; plasma renin activity; renin angiotensin aldosterone system; direct renin inhibitors; BNP; KCCQ; eGFR; (NYHA class II to IV) with elevated; BNP and reduced LVEF
MeSH Terms: interventions — Enalapril; aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combination Aliskiren / Enalapril (Experimental): Aliskiren / Enalapril combination therapy-150 mg/10 mg titrated to 300 mg/ 10 mg film-coated tablets and administered orally.
  Interventions: Drug: Enalapril; Drug: Aliskiren
- Aliskiren (Experimental): Aliskiren monotherapy - 150 mg titrated to 300 mg film-coated tablets and administered orally.
  Interventions: Drug: Aliskiren
- Enalapril (Active Comparator): Enalapril monotherapy -10 mg film-coated tablet and administered orally.
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Enalapril — Enalapril 10 mg film-coated tablet and administered orally.
  Arms: Combination Aliskiren / Enalapril; Enalapril
Drug: Aliskiren — Aliskiren 150 mg titrated to 300 mg film-coated tablet and administered orally.
  Other Names: SPP100
  Arms: Aliskiren; Combination Aliskiren / Enalapril

SUMMARY:
The study will evaluate the efficacy and safety of both aliskiren monotherapy and aliskiren/enalapril combination therapy as compared to enalapril monotherapy, on morbidity and mortality in patients with chronic heart failure (NYHA Class II - IV.

ELIGIBILITY:
Inclusion Criteria

Patients eligible for inclusion in this study had to fulfill all of the following criteria:

1. Patients ≥ 18 years of age, male or female.
2. Patients with a diagnosis of chronic heart failure (NYHA

   Class II - IV):
   1. LVEF ≤ 35% at Visit 1 (local measurement, within the past 6 months assessed by echocardiography, multiple uptake gated acquisition scan (MUGA), computerized tomography(CT) scan, magnetic resonance imaging (MRI) or ventricular angiography)
   2. Elevated BNP or NT-proBNP at Visit 1:

   BNP ≥ 150 pg/mL (or BNP ≥ 100 pg/mL and unplanned hospitalization for HF within the last 12 months prior to Visit 1) (according to local measurement). OR NT-proBNP ≥ 600 pg/mL (or NT-proBNP ≥ 400 pg/mL and unplanned hospitalization for HF within the last 12 months prior to Visit 1) (according to local measurement).
3. Patients had to be treated with an ACEI at a stable dose enalapril 10 mg daily at least or any other ACEI, e.g. ramipril, quinapril, lisinopril, fosinopril, perindopril, trandolapril; based on equivalent doses, for at least 4 weeks prior to Visit 1
4. Patients had to be treated with a beta-blocker, unless contraindicated or not tolerated, at a stable dose for at least 4 weeks prior to visit 1 (for patients not on target dose, according to local guidelines, or in absence of that medication, the reason should be documented).
5. Written informed consent to participate in the study and ability to comply with all requirements.

Exclusion Criteria

Patients with any of the following were to be excluded from participation in the study:

1. History of hypersensitivity to any of the study drugs including history or allergy to ACEIs as well as known or suspected contraindications to the study drugs or previous history of intolerance to high doses of ACEIs during up- titration process.
2. Patients treated concomitantly with both an ARB and an aldosterone antagonist in addition to study drug at Visit 1.
3. Current acute decompensated HF (defined as an acute exacerbation of a chronic heart failure status manifested by typical signs and symptoms of HF like dyspnea, fatigue etc., that may require IV therapy with diuretics, vasodilators and/or inotropic drugs).
4. Symptomatic hypotension and/or less than 95 mmHg systolic blood pressure (SBP) at Visit 1 and/or less than 90 mmHg SBP at Visit 4.
5. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or major vascular surgery, percutaneous coronary intervention (PCI) or carotid angioplasty, within the past 3 months prior to Visit 1.
6. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 6 months after Visit 1.
7. Right heart failure due to severe pulmonary disease.
8. Patients with Diabetes Mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7064 (Actual)
Dates: Start 2009-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (643):
- United States (54):
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Pine Bluff, Arkansas
  - Novartis Investigative Site, Searcy, Arkansas
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, French Camp, California
  - Novartis Investigative Site, Inglewood, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Modesto, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Westlake Village, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Littleton, Colorado
  - Novartis Investigative Site, Boynton Beach, Florida
  - Novartis Investigative Site, Daytona Beach, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville Beach, Florida
  - Novartis Investigative Site, Miami Lakes, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Wellington, Florida
  - Novartis Investigative Site, Athens, Georgia
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Gillespie, Illinois
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Auburn, Maine
  - Novartis Investigative Site, Southfield, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Elmer, New Jersey
  - Novartis Investigative Site, Laurelton, New York
  - Novartis Investigative Site, Stony Brook, New York
  - Novartis Investigative Site, Wiliamsville, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Varnville, South Carolina
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Everett, Washington
  - Novartis Investigative Site, Kirkland, Washington
- Argentina (18):
  - Novartis Investigative Site, Bahía Blanca, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Coronel Suárez, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, San Isidro, Buenos Aires
  - Novartis Investigative Site, San Nicolás de los Arroyos, Buenos Aires
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Va Allende, Córdoba Province
  - Novartis Investigative Site, Villa María, Córdoba Province
  - Novartis Investigative Site, Posadas, Misiones Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Australia (11):
  - Novartis Investigative Site, Canberra, Australian Capital Territory
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Wollongong, New South Wales
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Launceston, Tasmania
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Prahran, Victoria
- Austria (5):
  - Novartis Investigative Site, Graz, Austria
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (12):
  - Novartis Investigative Site, Brussels, Belgium
  - Novartis Investigative Site, Anderlecht
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, De Pinte
  - Novartis Investigative Site, Eupen
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Ieper
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Turnhout
- Brazil (15):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Campina Grande do Sul, Paraná
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Londrina, Paraná
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Caxias do Sul, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Marília, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Tatuí, São Paulo
- Canada (9):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Saint John, New Brunswick
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Joliette, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
- China (19):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Baotou
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Xi'an
- Colombia (10):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Baranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Cartagena, Departamento de Bolívar
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Florida Blanca
  - Novartis Investigative Site, Medellín
- Costa Rica (3):
  - Novartis Investigative Site, Alajuela, Costa Rica
  - Novartis Investigative Site, San José, Costa Rica
  - Novartis Investigative Site, Guadalupe, San Jose, Costa Rica
- Czechia (15):
  - Novartis Investigative Site, Benešov, Czech Republic
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Český Krumlov, Czech Republic
  - Novartis Investigative Site, Jindřichův Hradec, Czech Republic
  - Novartis Investigative Site, Kolín, Czech Republic
  - Novartis Investigative Site, Kroměříž, Czech Republic
  - Novartis Investigative Site, Louny, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Pilsen, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Vyškov, Czech Republic
  - Novartis Investigative Site, Mariánské Lázně
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Pribram VIII
- Denmark (22):
  - Novartis Investigative Site, Aalborg, Denmark
  - Novartis Investigative Site, Hellerup, Denmark
  - Novartis Investigative Site, Hvidovre, Denmark
  - Novartis Investigative Site, Silkeborg, Denmark
  - Novartis Investigative Site, Århus N
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Copenhagen S
  - Novartis Investigative Site, Elsinore
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Fredericia
  - Novartis Investigative Site, Frederiksberg
  - Novartis Investigative Site, Glostrup Municipality
  - Novartis Investigative Site, Hillerød
  - Novartis Investigative Site, Hjørring
  - Novartis Investigative Site, Holbæk
  - Novartis Investigative Site, Køge
  - Novartis Investigative Site, Næstved
  - Novartis Investigative Site, Odense C
  - Novartis Investigative Site, Randers NØ
  - Novartis Investigative Site, Svendborg
  - Novartis Investigative Site, Viborg
- Dominican Republic (2):
  - Novartis Investigative Site, Santo Domingo, Republica Dominicana
  - Novartis Investigative Site, San Cristóbal, San Cristóbal
- Estonia (4):
  - Novartis Investigative Site, Tallinn, Estonia
  - Novartis Investigative Site, Pärnu
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (5):
  - Novartis Investigative Site, Seinäjoki, Finland
  - Novartis Investigative Site, Ekenäs
  - Novartis Investigative Site, Hyvinkää
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Turku
- France (11):
  - Novartis Investigative Site, Albi
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bécon-les-Granits
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Saint-Etienne
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (78):
  - Novartis Investigative Site, Göttingen, Germany
  - Novartis Investigative Site, Winsen, Lower Saxony
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Nauheim
  - Novartis Investigative Site, Bad Neustadt an der Saale
  - Novartis Investigative Site, Bensheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Brake
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dinkelsbühl
  - Novartis Investigative Site, Dorsten
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Ebersbach
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Erkner
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gotha
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Gütersloh
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Haßloch
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Helmbrechts
  - Novartis Investigative Site, Heppenheim an der Bergstrasse
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kleve
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Königsbrück
  - Novartis Investigative Site, Köthen
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Lambrecht
  - Novartis Investigative Site, Landshut
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lichtentanne
  - Novartis Investigative Site, Lienen
  - Novartis Investigative Site, Loerrach
  - Novartis Investigative Site, Ludwigsburg
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Markkleeberg
  - Novartis Investigative Site, Mayen
  - Novartis Investigative Site, Melsungen
  - Novartis Investigative Site, Muehldorf Am Inn
  - Novartis Investigative Site, Muehlheim An Der Ruhr
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Northeim
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Oelde
  - Novartis Investigative Site, Pirna
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Salzwedel
  - Novartis Investigative Site, Schwalmstadt
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Solingen
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Wedel
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Würzburg
  - Novartis Investigative Site, Zwickau
- Greece (6):
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chios
  - Novartis Investigative Site, Edessa
- India (25):
  - Novartis Investigative Site, Guntur, Andhra Pradesh
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Secunderabad, Andhra Pradesh
  - Novartis Investigative Site, Vijayawada, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Lucknow, India
  - Novartis Investigative Site, Mumbai, India
  - Novartis Investigative Site, Noida, India
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Delhi, New Delhi
  - Novartis Investigative Site, New Delhi, New Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Hyderabad
- Ireland (3):
  - Novartis Investigative Site, Co Dublin, Ireland
  - Novartis Investigative Site, Galway, Ireland
  - Novartis Investigative Site, Dublin
- Italy (44):
  - Novartis Investigative Site, Montescano, (pv)
  - Novartis Investigative Site, Pavia, (pv)
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Arezzo, AR
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Lumezzane, BS
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Cosenza, CS
  - Novartis Investigative Site, Forlì, FC
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Casarano, LE
  - Novartis Investigative Site, Cecina, LI
  - Novartis Investigative Site, Castelnuovo di Garfagnana, LU
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Passirana Di Rho, MI
  - Novartis Investigative Site, Pieve di Coriano, MN
  - Novartis Investigative Site, Massa, MS
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Cotignola, RA
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Rimini, RN
  - Novartis Investigative Site, Cava de' Tirreni, SA
  - Novartis Investigative Site, Poggibonsi, SI
  - Novartis Investigative Site, Sondalo, SO
  - Novartis Investigative Site, Sarzana, SP
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Vittorio Veneto, TV
  - Novartis Investigative Site, San Daniele del Friuli, UD
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Tradate, VA
  - Novartis Investigative Site, San Bonifacio, VR
- Japan (42):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Inba-gun, Chiba
  - Novartis Investigative Site, Chikushino-shi, Fukuoka
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Higashiibaraki-gun, Ibaraki
  - Novartis Investigative Site, Hitachi-Naka, Ibaraki
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokosuka, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Kita-ku, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Saga, Saga-ken
  - Novartis Investigative Site, Ureshino, Saga-ken
  - Novartis Investigative Site, Hamada, Shimane
  - Novartis Investigative Site, Komatsushimachō, Tokushima
  - Novartis Investigative Site, Tokushima, Tokushima
  - Novartis Investigative Site, Adachi-ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Hōfu, Yamaguchi
  - Novartis Investigative Site, Shūnan, Yamaguchi
  - Novartis Investigative Site, Ube, Yamaguchi
- Latvia (2):
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Lithuania (4):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius
- Mexico (7):
  - Novartis Investigative Site, Aguascalientes, Aguascalientes
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Querétaro City, Querétaro
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
  - Novartis Investigative Site, Culiacán, Sinaloa
- Netherlands (17):
  - Novartis Investigative Site, Enschede, Netherlands
  - Novartis Investigative Site, Zutphen, Netherlands
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Apeldoorn
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Dirksland
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Haarlem
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Leiderdorp
  - Novartis Investigative Site, Meppel
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Venlo
  - Novartis Investigative Site, Wildervank
  - Novartis Investigative Site, Zwolle
- Norway (3):
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Trondheim
  - Novartis Investigative Site, Tønsberg
- Peru (10):
  - Novartis Investigative Site, Trujillo, La Libertad
  - Novartis Investigative Site, Chiclayo, Lambayeque
  - Novartis Investigative Site, Lima, Lima Province
  - Novartis Investigative Site, Bellavista, Lima region
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, Miraflores, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Juan de Miraflores, Lima region
- Poland (23):
  - Novartis Investigative Site, Bytom
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Gliwice
  - Novartis Investigative Site, Grodzisk Mazowiecki
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Kłodzko
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Ostrowiec Świętokrzyski
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Oława
  - Novartis Investigative Site, Piotrkow Trybunalski
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Płock
  - Novartis Investigative Site, Sandomierz
  - Novartis Investigative Site, Tarnów
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zabrze
  - Novartis Investigative Site, Łomża
- Portugal (8):
  - Novartis Investigative Site, Amadora, Portugal
  - Novartis Investigative Site, Carnaxide, Portugal
  - Novartis Investigative Site, Coimbra, Portugal
  - Novartis Investigative Site, Lisbon, Portugal
  - Novartis Investigative Site, Penafiel, Portugal
  - Novartis Investigative Site, Porto, Portugal
  - Novartis Investigative Site, Aveiro
  - Novartis Investigative Site, Faro
- Puerto Rico (3):
  - Novartis Investigative Site, Humacao
  - Novartis Investigative Site, Ponce
  - Novartis Investigative Site, San Juan
- Romania (15):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Iași, Jud Iasi
  - Novartis Investigative Site, Târgu Mureş, Jud Mures
  - Novartis Investigative Site, Iași, Jud. Iasi
  - Novartis Investigative Site, Târgu Mureş, Mureș County
  - Novartis Investigative Site, Brasov, Romania
  - Novartis Investigative Site, Oradea, Romania
  - Novartis Investigative Site, Timișoara, Romania
  - Novartis Investigative Site, Baia Mare
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Iași
  - Novartis Investigative Site, Piteşti
  - Novartis Investigative Site, Târgu Mureş
  - Novartis Investigative Site, Timișoara
- Russia (22):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Kursk
  - Novartis Investigative Site, Lyubertsy
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Pushkin,St-Petersburg
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Volgograd
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (18):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Komárno, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Levice, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Považská Bystrica, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Stropkov, Slovak Republic
  - Novartis Investigative Site, Žilina, Slovak Republic
  - Novartis Investigative Site, Bardejov, Slovakia
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Lučenec, Slovakia
  - Novartis Investigative Site, Prešov, Slovakia
  - Novartis Investigative Site, Trebišov, Slovakia
  - Novartis Investigative Site, Trenčín, Slovakia
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Piešťany
  - Novartis Investigative Site, Žilina
- South Africa (7):
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Benoni
  - Novartis Investigative Site, Boksburg
  - Novartis Investigative Site, Centurion
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Western Cape
  - Novartis Investigative Site, Worcester
- South Korea (8):
  - Novartis Investigative Site, Gwangju, Gwangju
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Spain (17):
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Utrera, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Tortosa, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Valdemoro, Madrid
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
- Sweden (16):
  - Novartis Investigative Site, Malmo, Sweden
  - Novartis Investigative Site, Nässjö, Sweden
  - Novartis Investigative Site, Falun
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Karlstad
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Mölndal
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Skellefteå
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Sundsvall
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Västerås
- Switzerland (9):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bellinzona
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Biel
  - Novartis Investigative Site, Bruderholz
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Olten
  - Novartis Investigative Site, Winterthur
  - Novartis Investigative Site, Zurich
- Taiwan (7):
  - Novartis Investigative Site, Yongkang District, Tainan
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Linkou District
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (10):
  - Novartis Investigative Site, Aydin, Turkey
  - Novartis Investigative Site, Istanbul, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Balcova / Izmir
  - Novartis Investigative Site, Etlik / Ankara
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Kinikli / Denizli
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Sivas
- United Kingdom (15):
  - Novartis Investigative Site, Leicester, Leicestershire
  - Novartis Investigative Site, Dafen, Llanelli
  - Novartis Investigative Site, Addlestone, Surrey
  - Novartis Investigative Site, Chichester, West Sussex
  - Novartis Investigative Site, Worthing, West Sussex
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Chesterfield
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Swindon
- Venezuela (7):
  - Novartis Investigative Site, Barcelona, Anzoátegui
  - Novartis Investigative Site, Puerto Ordaz and San Felix, Bolívar
  - Novartis Investigative Site, Caracas, Distrito Federal
  - Novartis Investigative Site, Valencia, Edo. Carabobo
  - Novartis Investigative Site, Caracas, Miranda
  - Novartis Investigative Site, Cumaná, Sucre
  - Novartis Investigative Site, Maracaibo, Zulia

REFERENCES:
- [Derived] Patel-Murray NL, Zhang L, Claggett BL, Xu D, Serrano-Fernandez P, Healey M, Wandel S, Chen CW, Jacob J, Xu H, Turner GM, Chutkow W, Yates DP, O'Donnell CJ, Prescott MF, Lefkowitz M, Gimpelewicz CR, Beste MT, Zhao F, Gou L, Desai AS, Jhund PS, Packer M, Pfeffer MA, Redfield MM, Rouleau JL, Zannad F, Zile MR, McMurray JJV, Mendelson MM, Solomon SD, Cunningham JW. Aptamer Proteomics for Biomarker Discovery in Heart Failure With Preserved Ejection Fraction: The PARAGON-HF Proteomic Substudy. J Am Heart Assoc. 2024 Jul 2;13(13):e033544. doi: 10.1161/JAHA.123.033544. Epub 2024 Jun 21. PMID 38904251
- [Derived] Kondo T, Dewan P, Anand IS, Desai AS, Packer M, Zile MR, Pfeffer MA, Solomon SD, Abraham WT, Shah SJ, Lam CSP, Jhund PS, McMurray JJV. Clinical Characteristics and Outcomes in Patients With Heart Failure: Are There Thresholds and Inflection Points in Left Ventricular Ejection Fraction and Thresholds Justifying a Clinical Classification? Circulation. 2023 Aug 29;148(9):732-749. doi: 10.1161/CIRCULATIONAHA.122.063642. Epub 2023 Jun 27. PMID 37366061
- [Derived] Shen L, Claggett BL, Jhund PS, Abraham WT, Desai AS, Dickstein K, Gong J, Kober LV, Lefkowitz MP, Rouleau JL, Shi VC, Swedberg K, Zile MR, Solomon SD, McMurray JJV. Development and external validation of prognostic models to predict sudden and pump-failure death in patients with HFrEF from PARADIGM-HF and ATMOSPHERE. Clin Res Cardiol. 2021 Aug;110(8):1334-1349. doi: 10.1007/s00392-021-01888-x. Epub 2021 Jun 8. PMID 34101002
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502
- [Derived] Kristensen SL, Castagno D, Shen L, Jhund PS, Docherty KF, Rorth R, Abraham WT, Desai AS, Dickstein K, Rouleau JL, Zile MR, Swedberg K, Packer M, Solomon SD, Kober L, McMurray JJV; PARADIGM-HF and ATMOSPHERE Committees and Investigators.. Prevalence and incidence of intra-ventricular conduction delays and outcomes in patients with heart failure and reduced ejection fraction: insights from PARADIGM-HF and ATMOSPHERE. Eur J Heart Fail. 2020 Dec;22(12):2370-2379. doi: 10.1002/ejhf.1972. Epub 2020 Sep 14. PMID 32720404
- [Derived] Docherty KF, Shen L, Castagno D, Petrie MC, Abraham WT, Bohm M, Desai AS, Dickstein K, Kober LV, Packer M, Rouleau JL, Solomon SD, Swedberg K, Vazir A, Zile MR, Jhund PS, McMurray JJV. Relationship between heart rate and outcomes in patients in sinus rhythm or atrial fibrillation with heart failure and reduced ejection fraction. Eur J Heart Fail. 2020 Mar;22(3):528-538. doi: 10.1002/ejhf.1682. Epub 2019 Dec 17. PMID 31849164
- [Derived] Dewan P, Rorth R, Raparelli V, Campbell RT, Shen L, Jhund PS, Petrie MC, Anand IS, Carson PE, Desai AS, Granger CB, Kober L, Komajda M, McKelvie RS, O'Meara E, Pfeffer MA, Pitt B, Solomon SD, Swedberg K, Zile MR, McMurray JJV. Sex-Related Differences in Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2019 Dec;12(12):e006539. doi: 10.1161/CIRCHEARTFAILURE.119.006539. Epub 2019 Dec 9. PMID 31813280
- [Derived] Shen L, Ramires F, Martinez F, Bodanese LC, Echeverria LE, Gomez EA, Abraham WT, Dickstein K, Kober L, Packer M, Rouleau JL, Solomon SD, Swedberg K, Zile MR, Jhund PS, Gimpelewicz CR, McMurray JJV; PARADIGM-HF and ATMOSPHERE Investigators and Committees. Contemporary Characteristics and Outcomes in Chagasic Heart Failure Compared With Other Nonischemic and Ischemic Cardiomyopathy. Circ Heart Fail. 2017 Nov;10(11):e004361. doi: 10.1161/CIRCHEARTFAILURE.117.004361. PMID 29141857
- [Derived] Kristensen SL, Jhund PS, Mogensen UM, Rorth R, Abraham WT, Desai A, Dickstein K, Rouleau JL, Zile MR, Swedberg K, Packer M, Solomon SD, Kober L, McMurray JJV; PARADIGM-HF and ATMOSPHERE Committees and Investigators. Prognostic Value of N-Terminal Pro-B-Type Natriuretic Peptide Levels in Heart Failure Patients With and Without Atrial Fibrillation. Circ Heart Fail. 2017 Oct;10(10):e004409. doi: 10.1161/CIRCHEARTFAILURE.117.004409. PMID 29018174
- [Derived] Kristensen SL, Mogensen UM, Tarnesby G, Gimpelewicz CR, Ali MA, Shao Q, Chiang Y, Jhund PS, Abraham WT, Dickstein K, McMurray JJV, Kober L. Aliskiren alone or in combination with enalapril vs. enalapril among patients with chronic heart failure with and without diabetes: a subgroup analysis from the ATMOSPHERE trial. Eur J Heart Fail. 2018 Jan;20(1):136-147. doi: 10.1002/ejhf.896. Epub 2017 Sep 25. PMID 28948656
- [Derived] McMurray JJ, Krum H, Abraham WT, Dickstein K, Kober LV, Desai AS, Solomon SD, Greenlaw N, Ali MA, Chiang Y, Shao Q, Tarnesby G, Massie BM; ATMOSPHERE Committees Investigators. Aliskiren, Enalapril, or Aliskiren and Enalapril in Heart Failure. N Engl J Med. 2016 Apr 21;374(16):1521-32. doi: 10.1056/NEJMoa1514859. Epub 2016 Apr 4. PMID 27043774

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During Active Run-in period, patients received enalapril for step 1 & 2 and then aliskiren on top of the max tolerated dose of enalapril for step 3. Patients who completed the run in were randomized in a 1:1:1 ratio to one of the 3 treatment arms (aliskiren/enalapril combination therapy, aliskiren monotherapy, or enalapril monotherapy).
Period: Overall Study
Arm/Group | Combination Aliskiren / Enalapril | Aliskiren | Enalapril
Started | 2354 | 2356 | 2354
Full Analysis Set (FAS) | 2340 | 2340 | 2336
Safety Set | 2347 | 2348 | 2345
Completed | 1567 | 1524 | 1539
Not Completed | 787 | 832 | 815
Not completed — Death | 713 | 768 | 753
Not completed — Lost to Follow-up | 11 | 6 | 11
Not completed — H.A. Request | 26 | 23 | 19
Not completed — IRB request | 0 | 0 | 2
Not completed — Vital Status known (alive) at study end | 2 | 3 | 3
Not completed — Vital Status unknown at study end | 1 | 1 | 0
Not completed — Vital Status at study end N/A | 8 | 10 | 10
Not completed — Patient's request | 21 | 17 | 11
Not completed — Missing study completion information | 5 | 4 | 6

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) - included all randomized patients but excluded 48 patients (22 mis-randomized but took no double blind and 26 patients due to GCP violations)
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Aliskiren / Enalapril | Aliskiren | Enalapril | Total
Number analyzed (Participants) | 2340 | 2340 | 2336 | 7016
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.65) | 63.3 (12.06) | 63.3 (11.71) | 63.2 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494 | 532 | 499 | 1525
  Male | 1846 | 1808 | 1837 | 5491

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had First Occurrence of the Composite Endpoint, Which is Defined as Either Cardiovascular (CV) Death or Heart Failure (HF) Hospitalization
Description: Number of participants that had first occurrence of the composite endpoint, which is defined as either CV death or HF hospitalization due to HF.
Time Frame: up to End of Study (78 months)
Population: Full Analysis Set (FAS) - All randomized patients with exception of mis-randomized patients that took no study drug and patients from the sites with major GCP violations.
Measure: Number; unit: participants
Arm/Group | Combination Aliskiren / Enalapril | Aliskiren | Enalapril
Number analyzed (Participants) | 2340 | 2340 | 2336
participants
  Primary Composite | 770 | 791 | 808
  CV death | 512 | 562 | 547
  1st HF Hospitalization | 430 | 442 | 452
Statistical Analysis 1: Comparison: Combination Aliskiren / Enalapril vs Enalapril; (superiority); Test type: Superiority or Other; p = 0.1724, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.85 to 1.03]
Statistical Analysis 2: Comparison: Combination Aliskiren / Enalapril vs Enalapril; (superiority) Non-Diabetic patients; Test type: Superiority or Other; p = 0.4579, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.85 to 1.07]
Statistical Analysis 3: Comparison: Aliskiren vs Enalapril; Test type: Non-Inferiority or Equivalence — Pre-specified Non-inferiority margin 1.104 is used; p = 0.0368, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.90 to 1.10]
Statistical Analysis 4: Comparison: Aliskiren vs Enalapril; (superiority); Test type: Superiority or Other; p = 0.9118, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.90 to 1.10]

2. Secondary Outcome: Change From Baseline to Month 12 for the Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score
Description: Change from baseline to Month 12 for the Kansas City Cardiomyopathy Questionnaire (KCCQ) clinical summary score. KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. KCCQ clinical summary score is a composite assessment of physical limitations and total symptom scores. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: KCCQ Score
Arm/Group | Combination Aliskiren / Enalapril | Aliskiren | Enalapril
Number analyzed (Participants) | 2340 | 2340 | 2336
KCCQ Score | -5.04 (0.56) | -6.03 (0.57) | -5.01 (0.55)

3. Secondary Outcome: All Cause Death
Description: Number of patients - All-cause death. All-cause death is common in Heart Failure HF patients this measures how many patients had this event.
Time Frame: up to end of study (78 months)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combination Aliskiren / Enalapril | Aliskiren | Enalapril
Number analyzed (Participants) | 2340 | 2340 | 2336
participants | 595 | 654 | 646

ADVERSE EVENTS:
Description: Safety set (SAF) (double-blind phase) - All patients who received at least one dose of double-blind study drug. Patients were analyzed according to treatment received.
  Treatment received was considered identical to the randomized treatment if the patient had received at least one dose of the randomized treatment.
Groups:
- Combination of Aliskiren and Enalapril: Aliskiren/Enalapril combination therapy-150 mg/10 mg titrated to 300 mg/ 10 mg
Arm/Group | Combination of Aliskiren and Enalapril | Aliskiren | Enalapril
Serious Adverse Events (participants affected / at risk) | 1466/2347 | 1504/2348 | 1501/2345
Other Adverse Events (participants affected / at risk) | 1698/2347 | 1605/2348 | 1623/2345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Aliskiren and Enalapril (N=2347) | Aliskiren (N=2348) | Enalapril (N=2345)
Acquired haemophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 36 | 28 | 28
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 | 0 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Bone marrow infiltration (Blood and lymphatic system disorders) | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypocoagulable state (Blood and lymphatic system disorders) | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Jaundice acholuric (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 4 | 2 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Splenic embolism (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 2 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 3
Acute coronary syndrome (Cardiac disorders) | 6 | 18 | 16
Acute left ventricular failure (Cardiac disorders) | 3 | 5 | 9
Acute myocardial infarction (Cardiac disorders) | 49 | 40 | 46
Adams-Stokes syndrome (Cardiac disorders) | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 35 | 33 | 37
Angina unstable (Cardiac disorders) | 47 | 48 | 41
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 3 | 1 | 3
Aortic valve stenosis (Cardiac disorders) | 3 | 3 | 1
Arrhythmia (Cardiac disorders) | 13 | 15 | 12
Arrhythmia supraventricular (Cardiac disorders) | 0 | 2 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 4 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 89 | 98 | 97
Atrial flutter (Cardiac disorders) | 15 | 21 | 11
Atrial tachycardia (Cardiac disorders) | 1 | 4 | 2
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 2
Atrioventricular block (Cardiac disorders) | 1 | 1 | 3
Atrioventricular block complete (Cardiac disorders) | 7 | 8 | 13
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 3 | 4 | 6
Bifascicular block (Cardiac disorders) | 1 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 3 | 2
Bradycardia (Cardiac disorders) | 12 | 12 | 9
Bundle branch block (Cardiac disorders) | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 4 | 4 | 3
Cardiac aneurysm (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 59 | 61 | 59
Cardiac asthma (Cardiac disorders) | 2 | 4 | 1
Cardiac discomfort (Cardiac disorders) | 3 | 3 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 480 | 521 | 503
Cardiac failure acute (Cardiac disorders) | 54 | 43 | 60
Cardiac failure chronic (Cardiac disorders) | 120 | 125 | 122
Cardiac failure congestive (Cardiac disorders) | 76 | 85 | 79
Cardiac flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac hypertrophy (Cardiac disorders) | 0 | 1 | 0
Cardiac perforation (Cardiac disorders) | 0 | 1 | 0
Cardiac sarcoidosis (Cardiac disorders) | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 2
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 24 | 24 | 20
Cardiogenic shock (Cardiac disorders) | 31 | 49 | 38
Cardiomegaly (Cardiac disorders) | 0 | 2 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 2 | 4
Cardiopulmonary failure (Cardiac disorders) | 4 | 6 | 2
Cardiorenal syndrome (Cardiac disorders) | 2 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 2
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 1
Chordae tendinae rupture (Cardiac disorders) | 0 | 0 | 1
Chronotropic incompetence (Cardiac disorders) | 0 | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 14 | 14 | 19
Coronary artery disease (Cardiac disorders) | 28 | 27 | 22
Coronary artery insufficiency (Cardiac disorders) | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 8 | 5 | 8
Coronary artery thrombosis (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Heart valve incompetence (Cardiac disorders) | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 2 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 13 | 7 | 13
Left ventricular dysfunction (Cardiac disorders) | 6 | 6 | 8
Left ventricular failure (Cardiac disorders) | 6 | 5 | 6
Metabolic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 6 | 17 | 14
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 56 | 50 | 50
Myocardial ischaemia (Cardiac disorders) | 19 | 19 | 18
Nodal rhythm (Cardiac disorders) | 1 | 1 | 0
Palpitations (Cardiac disorders) | 2 | 1 | 1
Papillary muscle rupture (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 3 | 2
Pericarditis (Cardiac disorders) | 1 | 0 | 1
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 1 | 3
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Rhythm idioventricular (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 2 | 1 | 2
Sinoatrial block (Cardiac disorders) | 1 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 6 | 3 | 5
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 2 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 7 | 5 | 3
Systolic dysfunction (Cardiac disorders) | 1 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 9 | 5 | 4
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 3 | 2
Ventricular arrhythmia (Cardiac disorders) | 14 | 8 | 14
Ventricular dysfunction (Cardiac disorders) | 0 | 2 | 2
Ventricular dyssynchrony (Cardiac disorders) | 2 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 8 | 9 | 3
Ventricular failure (Cardiac disorders) | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 32 | 30 | 34
Ventricular flutter (Cardiac disorders) | 2 | 2 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 2 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 78 | 67 | 63
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 3
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 1 | 1
Haematotympanum (Ear and labyrinth disorders) | 1 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 3 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 2 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 5 | 2
Hypothyroidism (Endocrine disorders) | 2 | 7 | 2
Thyrotoxic crisis (Endocrine disorders) | 1 | 0 | 0
Toxic nodular goitre (Endocrine disorders) | 0 | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0 | 0
Amblyopia (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 13 | 8 | 6
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1 | 1
Glaucoma (Eye disorders) | 0 | 1 | 1
Macular hole (Eye disorders) | 0 | 1 | 1
Ocular fistula (Eye disorders) | 0 | 0 | 1
Ocular retrobulbar haemorrhage (Eye disorders) | 1 | 0 | 0
Ophthalmic vein thrombosis (Eye disorders) | 0 | 0 | 1
Retinal artery embolism (Eye disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 0
Retinal degeneration (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 2
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 3 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 14 | 10 | 11
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 5 | 4
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Acid peptic disease (Gastrointestinal disorders) | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 1 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Anal prolapse (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 6 | 6 | 6
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1 | 3
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 5 | 2
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 4 | 11
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 2 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 2 | 5
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 3 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 2
Faecaloma (Gastrointestinal disorders) | 1 | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2 | 3
Gastric polyps (Gastrointestinal disorders) | 1 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 7 | 4 | 8
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 6 | 2 | 5
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 10 | 4 | 4
Gastritis erosive (Gastrointestinal disorders) | 1 | 1 | 3
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 19 | 13 | 11
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 4
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 4
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 4 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 5 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 2 | 0
Ileus (Gastrointestinal disorders) | 4 | 3 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 | 2 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 23 | 21 | 14
Intestinal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 4
Intestinal obstruction (Gastrointestinal disorders) | 2 | 3 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 1 | 3
Intestinal strangulation (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 2
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 2 | 5 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 4
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 1 | 0
Melaena (Gastrointestinal disorders) | 3 | 4 | 4
Mesenteric artery embolism (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 2 | 0 | 0
Mesenteritis (Gastrointestinal disorders) | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 4 | 3
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 2 | 2
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 5 | 4 | 2
Pancreatitis acute (Gastrointestinal disorders) | 9 | 5 | 5
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 7 | 5 | 3
Rectal polyp (Gastrointestinal disorders) | 1 | 1 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Stress ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 1
Tongue oedema (Gastrointestinal disorders) | 1 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 5 | 5 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 12 | 7
Visceral congestion (Gastrointestinal disorders) | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 1
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 5 | 4
Abasia (General disorders) | 0 | 2 | 0
Accidental death (General disorders) | 0 | 1 | 1
Asthenia (General disorders) | 8 | 5 | 4
Brain death (General disorders) | 0 | 0 | 1
Cardiac complication associated with device (General disorders) | 2 | 1 | 0
Cardiac death (General disorders) | 51 | 68 | 87
Chest discomfort (General disorders) | 2 | 0 | 0
Chest pain (General disorders) | 2 | 3 | 1
Death (General disorders) | 75 | 84 | 82
Device battery issue (General disorders) | 13 | 9 | 14
Device breakage (General disorders) | 1 | 0 | 1
Device defective (General disorders) | 0 | 0 | 1
Device dislocation (General disorders) | 1 | 4 | 2
Device electrical impedance issue (General disorders) | 2 | 0 | 0
Device end of service (General disorders) | 0 | 0 | 2
Device failure (General disorders) | 4 | 0 | 0
Device inappropriate shock delivery (General disorders) | 1 | 4 | 3
Device issue (General disorders) | 1 | 0 | 1
Device lead damage (General disorders) | 1 | 3 | 2
Device lead issue (General disorders) | 1 | 1 | 2
Device malfunction (General disorders) | 7 | 10 | 9
Device signal detection issue (General disorders) | 0 | 1 | 0
Device stimulation issue (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 5 | 1 | 2
Feeling abnormal (General disorders) | 1 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 3 | 3 | 7
Generalised oedema (General disorders) | 2 | 2 | 2
Hernia (General disorders) | 0 | 1 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 1 | 1
Implant site erosion (General disorders) | 0 | 0 | 1
Implant site haemorrhage (General disorders) | 1 | 0 | 0
Implant site necrosis (General disorders) | 0 | 1 | 0
Implant site pain (General disorders) | 0 | 0 | 1
Implant site ulcer (General disorders) | 1 | 0 | 0
Incarcerated hernia (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Injury associated with device (General disorders) | 0 | 0 | 1
Lead dislodgement (General disorders) | 1 | 1 | 1
Localised oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 5 | 4 | 1
Medical device complication (General disorders) | 4 | 1 | 1
Medical device site thrombosis (General disorders) | 0 | 0 | 1
Metaplasia (General disorders) | 1 | 1 | 0
Multi-organ failure (General disorders) | 21 | 15 | 12
Necrosis (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 13 | 15 | 22
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 9 | 6 | 3
Organ failure (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 5 | 8 | 7
Stent-graft endoleak (General disorders) | 0 | 1 | 0
Sudden cardiac death (General disorders) | 38 | 39 | 50
Sudden death (General disorders) | 98 | 89 | 86
Thrombosis in device (General disorders) | 0 | 0 | 1
Ulcer (General disorders) | 1 | 0 | 0
Ulcer haemorrhage (General disorders) | 0 | 1 | 1
Undersensing (General disorders) | 0 | 1 | 0
Vascular stent restenosis (General disorders) | 1 | 0 | 0
Vascular stent stenosis (General disorders) | 0 | 0 | 1
Vascular stent thrombosis (General disorders) | 0 | 1 | 2
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 2 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 3 | 3 | 0
Biliary cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 5 | 3
Cholangitis acute (Hepatobiliary disorders) | 2 | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 7 | 4 | 8
Cholecystitis acute (Hepatobiliary disorders) | 9 | 9 | 9
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 18 | 15 | 13
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Chronic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 2 | 6
Hepatic congestion (Hepatobiliary disorders) | 2 | 3 | 3
Hepatic failure (Hepatobiliary disorders) | 4 | 2 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 3 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 2 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 2 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 1 | 3
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 2 | 3 | 5
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 3 | 1
Jaundice hepatocellular (Hepatobiliary disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 1
Allergy to venom (Immune system disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Heart transplant rejection (Immune system disorders) | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 1 | 0
Abdominal sepsis (Infections and infestations) | 3 | 2 | 2
Abscess intestinal (Infections and infestations) | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 4
Abscess oral (Infections and infestations) | 0 | 1 | 0
Acinetobacter infection (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 3
Appendiceal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 5 | 2 | 5
Appendicitis perforated (Infections and infestations) | 2 | 2 | 2
Arthritis bacterial (Infections and infestations) | 1 | 3 | 1
Arthritis infective (Infections and infestations) | 2 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 2 | 1
Bacteraemia (Infections and infestations) | 1 | 1 | 1
Bacterial diarrhoea (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 1 | 1
Bacterial sepsis (Infections and infestations) | 1 | 1 | 2
Biliary sepsis (Infections and infestations) | 2 | 0 | 0
Bone abscess (Infections and infestations) | 0 | 1 | 0
Bone tuberculosis (Infections and infestations) | 0 | 0 | 1
Brain abscess (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 22 | 16 | 11
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1 | 1
Burn infection (Infections and infestations) | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 1
Cardiac valve abscess (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 6 | 9 | 13
Cholecystitis infective (Infections and infestations) | 3 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 1 | 0
Corynebacterium infection (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 6 | 1 | 3
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 6 | 6 | 4
Device related sepsis (Infections and infestations) | 0 | 3 | 0
Diabetic foot infection (Infections and infestations) | 3 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 6 | 0 | 4
Dysentery (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 1 | 1 | 0
Encephalitis (Infections and infestations) | 1 | 2 | 0
Endocarditis (Infections and infestations) | 5 | 5 | 4
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 0
Endocarditis staphylococcal (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 2 | 0
Erysipelas (Infections and infestations) | 6 | 7 | 10
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1
Fungal oesophagitis (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 10 | 3 | 2
Gastric ulcer helicobacter (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 13 | 10 | 16
Gastroenteritis clostridial (Infections and infestations) | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 2
Gastrointestinal infection (Infections and infestations) | 2 | 0 | 1
Genitourinary tract infection (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 2
H1N1 influenza (Infections and infestations) | 0 | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0 | 2
Haemophilus sepsis (Infections and infestations) | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Hepatic infection bacterial (Infections and infestations) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 4
Herpes zoster cutaneous disseminated (Infections and infestations) | 0 | 1 | 0
Human ehrlichiosis (Infections and infestations) | 1 | 0 | 0
Implant site infection (Infections and infestations) | 3 | 1 | 3
Incision site abscess (Infections and infestations) | 1 | 0 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 1
Infected seroma (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 2 | 4 | 3
Infection (Infections and infestations) | 4 | 2 | 4
Infectious colitis (Infections and infestations) | 1 | 1 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 2 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 4 | 2
Influenza (Infections and infestations) | 2 | 2 | 2
Intervertebral discitis (Infections and infestations) | 2 | 0 | 0
Intestinal sepsis (Infections and infestations) | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 5 | 4 | 3
Lower respiratory tract infection (Infections and infestations) | 5 | 6 | 9
Lung abscess (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 10 | 6 | 13
Lyme disease (Infections and infestations) | 0 | 0 | 1
Mucormycosis (Infections and infestations) | 0 | 0 | 1
Mycobacterial infection (Infections and infestations) | 0 | 1 | 0
Myiasis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 0
Necrotising fasciitis (Infections and infestations) | 2 | 1 | 2
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 1 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0
Orchitis (Infections and infestations) | 2 | 1 | 1
Oropharyngitis fungal (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 2
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 1
Parametritis (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 1
Peritonitis (Infections and infestations) | 2 | 3 | 6
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 2 | 5 | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 136 | 145 | 122
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 1 | 1
Post procedural sepsis (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 2 | 2
Prostatic abscess (Infections and infestations) | 0 | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 1
Psoas abscess (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 8 | 6 | 4
Pulmonary tuberculosis (Infections and infestations) | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 4 | 3 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 8 | 15 | 19
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection fungal (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 2 | 2
Sepsis (Infections and infestations) | 14 | 18 | 12
Septic necrosis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 13 | 21 | 13
Sialoadenitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 2 | 1 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Spinal cord infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 2 | 3
Streptococcal endocarditis (Infections and infestations) | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 3
Thrombophlebitis septic (Infections and infestations) | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 1 | 1
Tracheitis (Infections and infestations) | 1 | 1 | 0
Tracheobronchitis (Infections and infestations) | 6 | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 6
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Urethritis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 22 | 21 | 19
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 5 | 7 | 3
Viral infection (Infections and infestations) | 0 | 3 | 0
Viral pericarditis (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Viral vasculitis (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 2 | 1 | 1
Wound infection bacterial (Infections and infestations) | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Wound sepsis (Infections and infestations) | 1 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 4 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 3 | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 1 | 0
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 | 2 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 3 | 0
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Chest injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Closed globe injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Complications of transplanted heart (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 3 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 2 | 0
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 | 3 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 8 | 11
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 | 3 | 3
Femur fracture (Injury, poisoning and procedural complications) | 9 | 10 | 6
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 3 | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 2
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 7 | 3 | 3
Hip fracture (Injury, poisoning and procedural complications) | 4 | 5 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 2 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 2 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 4 | 9 | 0
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 2 | 3
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 3 | 2
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 4 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Product name confusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 5 | 5 | 1
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 8 | 6 | 8
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 3 | 2
Sacroiliac fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 4 | 2
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 5 | 5
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 6 | 3 | 3
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic shock (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Underdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 4 | 1
Urethral stricture traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 2 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1 | 0
Anticoagulation drug level increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 2
Blood creatinine increased (Investigations) | 7 | 4 | 5
Blood ethanol increased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 2
Blood magnesium decreased (Investigations) | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 2 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1
Blood urine (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1
Cardiac output decreased (Investigations) | 1 | 0 | 0
Cardioactive drug level increased (Investigations) | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 1 | 0
Coagulation test abnormal (Investigations) | 1 | 0 | 0
Coagulation time prolonged (Investigations) | 1 | 0 | 0
Ejection fraction abnormal (Investigations) | 1 | 2 | 1
Ejection fraction decreased (Investigations) | 1 | 0 | 1
Electrocardiogram QRS complex prolonged (Investigations) | 1 | 2 | 1
Enterobacter test positive (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 2
International normalised ratio abnormal (Investigations) | 1 | 1 | 0
International normalised ratio increased (Investigations) | 5 | 3 | 6
Lipase increased (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0
Viral load increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 3 | 3 | 1
Weight increased (Investigations) | 1 | 0 | 3
White blood cell count increased (Investigations) | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 3
Cachexia (Metabolism and nutrition disorders) | 1 | 1 | 0
Carbohydrate intolerance (Metabolism and nutrition disorders) | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 6 | 1
Dehydration (Metabolism and nutrition disorders) | 27 | 21 | 14
Diabetes mellitus (Metabolism and nutrition disorders) | 15 | 16 | 10
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 7 | 6 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 | 0 | 3
Fluid overload (Metabolism and nutrition disorders) | 3 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 11 | 11 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 21 | 13 | 20
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 5 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 12 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 7 | 10
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Insulin resistance (Metabolism and nutrition disorders) | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Marasmus (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0 | 2
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 1
Mineral deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 12 | 10 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 6 | 3 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 12 | 10
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 6
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8 | 2
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 3
Benign ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 6
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 3
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 7
Carcinoma in situ of penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 4 | 7
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3 | 3
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatobiliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 9 | 12
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 2
Malignant neoplasm of auricular cartilage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 7 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 3
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 5
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pineal parenchymal neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7 | 19
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 3
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 3
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Sinus cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 5
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ageusia (Nervous system disorders) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Atonic seizures (Nervous system disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Basilar artery stenosis (Nervous system disorders) | 0 | 1 | 0
Brain hypoxia (Nervous system disorders) | 0 | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 2 | 0
Brain stem infarction (Nervous system disorders) | 0 | 0 | 1
Brain stem syndrome (Nervous system disorders) | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 1 | 0
Carotid artery disease (Nervous system disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 5 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebellar ataxia (Nervous system disorders) | 1 | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 2 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral amyloid angiopathy (Nervous system disorders) | 0 | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0 | 5
Cerebral artery occlusion (Nervous system disorders) | 1 | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 0 | 2
Cerebral haematoma (Nervous system disorders) | 1 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 6 | 9 | 7
Cerebral infarction (Nervous system disorders) | 9 | 17 | 17
Cerebral ischaemia (Nervous system disorders) | 3 | 2 | 3
Cerebrovascular accident (Nervous system disorders) | 44 | 51 | 62
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0 | 0
Cervicogenic headache (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 2 | 1
Coma (Nervous system disorders) | 1 | 3 | 2
Complex partial seizures (Nervous system disorders) | 0 | 1 | 1
Dementia (Nervous system disorders) | 6 | 1 | 3
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 1
Diabetic coma (Nervous system disorders) | 0 | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 11 | 9 | 4
Dizziness postural (Nervous system disorders) | 1 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 1 | 3
Dyslalia (Nervous system disorders) | 0 | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 3 | 1 | 1
Encephalomalacia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 2 | 1
Epilepsy (Nervous system disorders) | 2 | 7 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 3 | 4 | 4
Headache (Nervous system disorders) | 1 | 3 | 1
Hemianopia (Nervous system disorders) | 0 | 0 | 1
Hemianopia homonymous (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 3 | 3 | 1
Hemiplegia (Nervous system disorders) | 0 | 2 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 2 | 0
Hydrocephalus (Nervous system disorders) | 2 | 0 | 2
Hypoglycaemic coma (Nervous system disorders) | 1 | 0 | 2
Hypoglycaemic seizure (Nervous system disorders) | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 | 2 | 3
IIIrd nerve paresis (Nervous system disorders) | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 2
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 45 | 45 | 29
Lacunar infarction (Nervous system disorders) | 1 | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 5 | 3 | 5
Mental retardation (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 2
Monoparesis (Nervous system disorders) | 1 | 1 | 1
Monoplegia (Nervous system disorders) | 0 | 0 | 2
Motor neurone disease (Nervous system disorders) | 1 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0
Narcolepsy (Nervous system disorders) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 2
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0 | 0
Paresis cranial nerve (Nervous system disorders) | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 2
Parkinsonism (Nervous system disorders) | 1 | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Postresuscitation encephalopathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 4 | 5 | 9
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1
Retrograde amnesia (Nervous system disorders) | 1 | 0 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 1 | 4 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 0 | 2 | 0
Spinal epidural haematoma (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 1 | 3
Syncope (Nervous system disorders) | 48 | 56 | 27
Tension headache (Nervous system disorders) | 0 | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 0 | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 23 | 20 | 15
Tremor (Nervous system disorders) | 1 | 1 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 1
Uraemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 2
Vascular dementia (Nervous system disorders) | 0 | 2 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 3 | 2 | 2
Abulia (Psychiatric disorders) | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 2 | 2
Anxiety (Psychiatric disorders) | 2 | 2 | 4
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1
Apathy (Psychiatric disorders) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Catatonia (Psychiatric disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 2 | 2
Confusional state (Psychiatric disorders) | 4 | 4 | 3
Delirium (Psychiatric disorders) | 1 | 3 | 2
Delusion (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 2 | 6 | 2
Disorientation (Psychiatric disorders) | 0 | 1 | 1
Fear (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 3 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0
Somatisation disorder (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 52 | 29 | 38
Acute prerenal failure (Renal and urinary disorders) | 1 | 2 | 2
Anuria (Renal and urinary disorders) | 1 | 1 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 2
Calculus ureteric (Renal and urinary disorders) | 1 | 2 | 1
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 21 | 10 | 10
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 6 | 5
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Ischaemic nephropathy (Renal and urinary disorders) | 1 | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 1 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 1
Polyuria (Renal and urinary disorders) | 2 | 1 | 0
Postrenal failure (Renal and urinary disorders) | 1 | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 1
Renal embolism (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 33 | 26 | 27
Renal impairment (Renal and urinary disorders) | 34 | 31 | 33
Renal infarct (Renal and urinary disorders) | 0 | 0 | 2
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0
Ureteric fistula (Renal and urinary disorders) | 0 | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 2
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 7 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2 | 0
Urinoma (Renal and urinary disorders) | 0 | 1 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 9 | 7
Breast hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Mammary fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 2
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0
Spermatocele (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 2 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 20 | 20 | 17
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 14
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 5
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 8
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 32 | 32 | 43
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 3
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 | 46 | 35
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 12
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Pleurocutaneous fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 | 18 | 9
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 4
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 27 | 27 | 14
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 | 16 | 26
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acquired epidermolysis bullosa (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 5 | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Fungating wound (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 4 | 4
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Immobile (Social circumstances) | 1 | 0 | 1
Treatment noncompliance (Social circumstances) | 0 | 1 | 0
Heart transplant (Surgical and medical procedures) | 0 | 1 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 3 | 1
Accelerated hypertension (Vascular disorders) | 5 | 1 | 1
Aneurysm ruptured (Vascular disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 8 | 8
Aortic aneurysm rupture (Vascular disorders) | 2 | 1 | 2
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Aortic dilatation (Vascular disorders) | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 2
Aortic rupture (Vascular disorders) | 0 | 2 | 0
Aortic stenosis (Vascular disorders) | 2 | 3 | 1
Aortic thrombosis (Vascular disorders) | 1 | 0 | 0
Arterial insufficiency (Vascular disorders) | 0 | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 3 | 1 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 0 | 1
Arteritis (Vascular disorders) | 1 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 7 | 3 | 3
Deep vein thrombosis (Vascular disorders) | 3 | 5 | 4
Diabetic vascular disorder (Vascular disorders) | 0 | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 1
Embolism venous (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 2 | 2 | 0
Femoral artery embolism (Vascular disorders) | 0 | 0 | 1
Femoral artery occlusion (Vascular disorders) | 2 | 3 | 2
Haematoma (Vascular disorders) | 5 | 1 | 4
Haemodynamic instability (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 17 | 13 | 10
Hypertensive crisis (Vascular disorders) | 7 | 4 | 3
Hypertensive emergency (Vascular disorders) | 2 | 0 | 1
Hypotension (Vascular disorders) | 37 | 49 | 26
Hypovolaemic shock (Vascular disorders) | 1 | 4 | 2
Iliac artery embolism (Vascular disorders) | 0 | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1 | 1
Intermittent claudication (Vascular disorders) | 5 | 5 | 3
Ischaemia (Vascular disorders) | 0 | 1 | 0
Ischaemic limb pain (Vascular disorders) | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 5 | 3 | 4
Peripheral arterial occlusive disease (Vascular disorders) | 18 | 13 | 11
Peripheral artery aneurysm (Vascular disorders) | 1 | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 5 | 2 | 3
Peripheral artery thrombosis (Vascular disorders) | 0 | 3 | 4
Peripheral embolism (Vascular disorders) | 4 | 2 | 3
Peripheral ischaemia (Vascular disorders) | 5 | 8 | 3
Peripheral vascular disorder (Vascular disorders) | 1 | 2 | 1
Peripheral venous disease (Vascular disorders) | 0 | 4 | 4
Post thrombotic syndrome (Vascular disorders) | 0 | 1 | 2
Secondary hypertension (Vascular disorders) | 1 | 0 | 0
Shock (Vascular disorders) | 2 | 1 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 1 | 2
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 2 | 1 | 2
Varicophlebitis (Vascular disorders) | 0 | 1 | 0
Varicose ulceration (Vascular disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 3 | 1
Vascular rupture (Vascular disorders) | 0 | 1 | 0
Venous haemorrhage (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Aliskiren and Enalapril (N=2347) | Aliskiren (N=2348) | Enalapril (N=2345)
Anaemia (Blood and lymphatic system disorders) | 124 | 115 | 111
Angina pectoris (Cardiac disorders) | 81 | 86 | 71
Atrial fibrillation (Cardiac disorders) | 199 | 238 | 184
Cardiac failure (Cardiac disorders) | 241 | 254 | 238
Ventricular tachycardia (Cardiac disorders) | 55 | 74 | 55
Constipation (Gastrointestinal disorders) | 96 | 79 | 82
Diarrhoea (Gastrointestinal disorders) | 145 | 117 | 116
Nausea (Gastrointestinal disorders) | 68 | 78 | 55
Fatigue (General disorders) | 96 | 107 | 101
Oedema peripheral (General disorders) | 182 | 183 | 176
Bronchitis (Infections and infestations) | 151 | 138 | 147
Influenza (Infections and infestations) | 91 | 62 | 86
Nasopharyngitis (Infections and infestations) | 185 | 187 | 186
Pneumonia (Infections and infestations) | 84 | 95 | 78
Upper respiratory tract infection (Infections and infestations) | 84 | 74 | 79
Urinary tract infection (Infections and infestations) | 92 | 82 | 84
Blood creatinine increased (Investigations) | 97 | 70 | 57
Glomerular filtration rate decreased (Investigations) | 88 | 50 | 79
Diabetes mellitus (Metabolism and nutrition disorders) | 99 | 96 | 84
Gout (Metabolism and nutrition disorders) | 113 | 88 | 91
Hyperkalaemia (Metabolism and nutrition disorders) | 469 | 283 | 350
Hyperuricaemia (Metabolism and nutrition disorders) | 101 | 108 | 93
Hypokalaemia (Metabolism and nutrition disorders) | 130 | 149 | 116
Arthralgia (Musculoskeletal and connective tissue disorders) | 72 | 86 | 71
Back pain (Musculoskeletal and connective tissue disorders) | 90 | 82 | 98
Dizziness (Nervous system disorders) | 179 | 140 | 144
Headache (Nervous system disorders) | 55 | 71 | 67
Insomnia (Psychiatric disorders) | 91 | 92 | 98
Renal impairment (Renal and urinary disorders) | 414 | 298 | 328
Cough (Respiratory, thoracic and mediastinal disorders) | 285 | 223 | 286
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 204 | 216 | 213
Hypertension (Vascular disorders) | 188 | 180 | 137
Hypotension (Vascular disorders) | 409 | 308 | 332

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.